CLINICAL TRIAL: NCT00183261
Title: A Randomized Phase II Study of Therapeutic Immunization and Treatment Interruption Among Subjects Who Began Potent Antiretroviral Therapy Within 30 Days of Diagnosis of Acute or Recent HIV Infection
Brief Title: Immune Response to a Therapeutic HIV Vaccine Followed by Treatment Interruption in Patients With Acute or Recent HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Acute Infection and Early Disease Research Program (Network); Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIN504/A5218; 10025 (Registry Identifier: DAIDS ES); AIN504/ACTG A5218; AIN504-A5218
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Treatment Interruption; HIV Therapeutic Vaccine; Acute Infection; Acute Retroviral Syndrome
MeSH Terms: conditions — HIV Infections; Acute Retroviral Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Experimental): Participants will receive the MRKAd5 HIV-1 gag/pol/nef vaccine at study entry and on Weeks 4 and 26
  Interventions: Biological: MRKAd5 HIV-1 gag/pol/nef
- 2 (Placebo Comparator): Participants will receive the MRKAd5 HIV-1 gag/pol/nef vaccine placebo at study entry and on Weeks 4 and 26
  Interventions: Biological: MRKAd5 HIV-1 gag/pol/nef placebo

INTERVENTIONS:
Biological: MRKAd5 HIV-1 gag/pol/nef — 1.5 x 1010 Ad vg/mL, 1.0 mL administered intramuscularly
  Arms: 1
Biological: MRKAd5 HIV-1 gag/pol/nef placebo — 1.0 mL administered intramuscularly
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the HIV vaccine MRKAd5 HIV-1 gag/pol/nef followed by treatment interruption can increase immune system function in adults with acute or recent HIV infection who have started taking anti-HIV drugs.

DETAILED DESCRIPTION:
While the advent of highly active antiretroviral therapy (HAART) has contributed to the increasing control of HIV infection and viral replication, ultimate control of HIV infection will require the development of effective HIV-specific immunity in HIV infected individuals. Therapeutic vaccination within the earliest weeks following acute or recent HIV infection may increase the immune system's response to HIV. This study will determine whether MRKAd5 HIV-1 gag/pol/nef vaccine followed by treatment interruption can maintain viral suppression in patients with acute or recent HIV infection.

The interventional part of the study will last 102 weeks. Participants will be randomly assigned to receive either MRKAd5 HIV-1 gag/pol/nef or placebo vaccine at baseline and Weeks 4 and 26. Participants must remain on HAART from study entry until Week 38. Participants whose HIV viral load rebounds two times or more above 500 copies/ml by Weeks 39 to 41 will not enter Step 2 of the study. Participants whose viral load drops to 500 copies/ml or less by Weeks 39 to 41 will enter Step 2, where they will discontinue HAART for 24 weeks. Participants in Step 2 will have plasma HIV viral loads measured every 2 weeks for the first 4 weeks and weekly for the next 3 weeks. Study participants will continue in Step 2 until they experience virologic and immunologic failure or they need to restart HAART for another reason; they will then enter Step 3, where they will reinitiate HAART. Step 3 participants will continue on HAART until Week 102. A long-term safety follow-up period will occur from Weeks 103 to 240.

Timing of the study visits will be determined by which steps a participant enters. A physical exam and blood and urine collection will occur at most study visits throughout the study until Week 102. Follow-up phone calls to study participants will occur every 6 months from Week 102 until Week 240 to collect long-term safety data, including clinical status, CD4 count, and medication history. During the long-term safety follow-up, participants will also have study visits every 6 months. Visits will include medical and medication history.

ELIGIBILITY:
Inclusion Criteria:

* Initiated HAART within 30 days of an acute or recent HIV-1 infection diagnosis. More information on this criterion can be found in the protocol.
* Initiated HAART within 30 days of documented acute or recent HIV-1 infection without interruption for more than 7 days
* Sustained viral suppression, defined as a viral load of 500 copies/mL or less 12 months prior to baseline with an undetectable HIV-1 RNA viral load between 60 to 7 days prior to baseline
* CD4 count of 450 cells/mm3 or more OR 35% or more between 60 to 14 days prior to baseline
* Ad5 neutralizing antibody titer of 200 or less at screening
* Willing to follow all study procedures and schedules
* Willing to interrupt HAART for at least 24 weeks following completion of the vaccination stage
* Negative for hepatitis B surface antigen (HBsAg) at screening
* Willing to use acceptable forms of contraception
* Infected with HIV-1 subtype B, if this information is available

Exclusion Criteria:

* Virologic relapse, defined as 2 consecutive measurements of viral load of 500 copies/mL or more at least 7 days apart within 12 months of baseline visit
* Received more than 7 days of continuous HAART other than that received within 16 days of acute or recent HIV-1 infection. Participants who received HAART as part of post-exposure prophylaxis (PEP) more than 6 months prior to the start of initial HAART may be eligible, provided that they did not acquire HIV-1 infection from the event that required PEP.
* History of anaphylaxis or allergy to vaccine components, including Tris buffer, magnesium chloride, and polysorbate 80 (Tween)
* History of clinically significant heart, lung, kidney, liver, pancreatic, gastrointestinal, or neurological disease that, in the opinion of the study investigator, may interfere with the study
* Contraindication to intramuscular (IM) injection, such as anticoagulant therapy or thrombocytopenia
* Receipt of any immune globulin or blood products within 3 months prior to baseline
* Receipt of any live vaccine within 30 days prior to baseline or any inactivated vaccine within 14 days prior to baseline
* Previous receipt of any HIV vaccine. Participants that were documented to have received only placebo are not excluded.
* History of any AIDS-defining illness. If a participant's sole AIDS-defining illness is Kaposi's sarcoma limited to the skin and is not anticipated to require systemic chemotherapy, that participant is not excluded.
* Currently receiving drugs or biologics not approved by the Food and Drug Administration (FDA) other than investigational HIV medications
* Current or past participation in other studies that might alter the participant's response to the study vaccination
* Use of any immunomodulatory agents, including but not limited to interleukin-2 (IL-2), granulocyte/macrophage-colony stimulating factor (GM-CSF), and systemic corticosteroids, within 30 days prior to baseline
* Active alcohol or substance use that, in the investigator's opinion, may interfere with the study
* Any other criteria or condition that, in the investigator's opinion, may interfere with the study
* Unwilling or unable to contribute to the planned peripheral blood mononuclear cell (PBMC) blood collection
* Pregnancy or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2006-03; Primary Completion 2007-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Average of log10 HIV-1 RNA viral load | At Weeks 58 and 63
Frequency of Grade 3 or 4 systemic adverse events, the occurrence of a severe or life-threatening injection site adverse event, or death | Throughout study

SECONDARY OUTCOMES:
Distribution of plasma HIV RNA viral load | At Weeks 63 and 87
Proportion of patients with controlled viremia and their respective distribution of plasma HIV RNA viral load | At Weeks 63 and 87
Mean viral burden, defined as time-averaged area under the log10 HIV-1 RNA viral load curve | At Weeks 63 and 87
HIV DNA levels | At Weeks 30, 38, 63, and 87
HIV-1 DNA levels | At Weeks 30, 38, 46, 50, 63, and 87
Magnitude and absolute change in CD4 and CD8 counts | At Weeks 63 and 87
Percent and absolute change in the number of HIV-1- specific CD8 cells, as measured by interferon (IFN)-gamma Elispot assay and intracellular cytokine staining | Through Week 30
Percent and absolute change in the cytokine secretion patterns and the proliferative capacity of HIV-1- specific CD4 and CD8 cells, as measured by multiparameter flow cytometry | Through Week 30
Breadth and magnitude of HIV-1- specific CD4 and CD8 cell responses | Throughout study
Time to reach the specified virologic or immunologic criteria for reinitiating antiretroviral therapy after treatment interruption | Throughout study
Frequency of Grade 3 or 4 systemic adverse events or the occurrence of a severe or life-threatening injection site adverse event, or HIV-related events, AIDS-defining infections, and death from time of vaccination | Throughout study
Cell-associated infectivity in latently infected cells | At Week 63
Cell-associated infectivity at Week 63 and immunologic responses | At Weeks 63 and 87

CONTACTS AND LOCATIONS:
Overall Officials: Susan Little, MD, Study Chair — University of California, San Diego AIDS Vaccine Research Center; Douglas D. Richman, MD, Study Chair — Departments of Pathology and Medicine, University of California, San Diego
Locations (23):
- United States (13):
  - Ucsd Aiedrp, San Diego, California
  - Ucsf Aiedrp, San Francisco, California
  - LA Biomedical Research Institute at Harbor-UCLA AIEDRP, Torrance, California
  - Univ. of Colorado Health Sciences Ctr. AIEDRP, Denver, Colorado
  - Fenway Community Health Ctr. CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Aaron Diamond AIDS Research Ctr. AIEDRP, New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - UNC, Chapel Hill AIEDRP, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Dumc Aiedrp, Durham, North Carolina
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
- 407 Doctors CRS, Surry Hills, New South Wales, American Samoa
- Australia (9):
  - Holdsworth House Medical Practice CRS, Darlinghurst, New South Wales
  - St. Vincent's Hospital CRS, Darlinghurst, New South Wales
  - Taylor Square Private Clinic CRS, Darlinghurst, New South Wales
  - AIDS Research Initiative, Darlinghurst CRS, Darlinghurst, New South Wales
  - 407 Doctors (Australia) AIEDRP, Sydney
  - AIDS Research Initiative (Australia) AIEDRP, Sydney
  - St. Vincent's Hosp. (Australia) AIEDRP, Sydney
  - Taylor Square Private Clinic (Australia) AIEDRP, Sydney
  - Holdsworth House Gen. Practice (Australia) AIEDRP, Sydney

REFERENCES:
- [Background] Markowitz M, Jin X, Hurley A, Simon V, Ramratnam B, Louie M, Deschenes GR, Ramanathan M Jr, Barsoum S, Vanderhoeven J, He T, Chung C, Murray J, Perelson AS, Zhang L, Ho DD. Discontinuation of antiretroviral therapy commenced early during the course of human immunodeficiency virus type 1 infection, with or without adjunctive vaccination. J Infect Dis. 2002 Sep 1;186(5):634-43. doi: 10.1086/342559. Epub 2002 Aug 9. PMID 12195350
- [Background] Moss RB, Brandt C, Giermakowska WK, Savary JR, Theofan G, Zanetti M, Carlo DJ, Wallace MR. HIV-specific immunity during structured antiviral drug treatment interruption. Vaccine. 2003 Mar 7;21(11-12):1066-71. doi: 10.1016/s0264-410x(02)00610-2. PMID 12559781
- [Background] Papasavvas E, Ortiz GM, Gross R, Sun J, Moore EC, Heymann JJ, Moonis M, Sandberg JK, Drohan LA, Gallagher B, Shull J, Nixon DF, Kostman JR, Montaner LJ. Enhancement of human immunodeficiency virus type 1-specific CD4 and CD8 T cell responses in chronically infected persons after temporary treatment interruption. J Infect Dis. 2000 Sep;182(3):766-75. doi: 10.1086/315748. Epub 2000 Aug 17. PMID 10950770
- [Background] Rosenberg ES, Altfeld M, Poon SH, Phillips MN, Wilkes BM, Eldridge RL, Robbins GK, D'Aquila RT, Goulder PJ, Walker BD. Immune control of HIV-1 after early treatment of acute infection. Nature. 2000 Sep 28;407(6803):523-6. doi: 10.1038/35035103. PMID 11029005